CLINICAL TRIAL: NCT05949099
Title: Phase II Study of Cryoablation and Nirogacestat for Desmoid Tumor
Brief Title: Study of Cryoablation and Nirogacestat for Desmoid Tumor
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nam Bui (Other)
Collaborators: SpringWorks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Nam Bui, Clinical Associate Professor, Medicine - Oncology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-67799; NCI-2023-05590 (Registry Identifier: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2023-07-07; First posted 2023-07-17 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Desmoid Tumor
Keywords: Desmoid; Cryoablation; Nirogacestat
MeSH Terms: conditions — Desmoid Tumors | interventions — nirogacestat; Cryosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nirogacestat 150 mg (Experimental): Patients will receive 3-cycle lead-in with systemic therapy with nirogacestat 150 mg po BID, given continuously.
  Interventions: Drug: Nirogacestat; Procedure: Cryoablation

INTERVENTIONS:
Drug: Nirogacestat — Nirogacestat 150 mg by mouth twice-daily continuously for Cycles 1 through 3. Treatment with nirogacestat may continue via this study protocol for up to 24 months (26 cycles of treatment), unless there is progression of disease, intolerance, start of new anticancer therapy, or Subject Study Completion or Termination occurs.
Procedure: Cryoablation — Cryoablation procedure (single session) of one tumor mass between Cycles 3 and 4 of nirogacestat treatment

SUMMARY:
The primary purpose of this protocol is Systemic therapy with oral study agent, nirogacestat, followed by a single cryoablation procedure.

DETAILED DESCRIPTION:
The primary purpose of this protocol is treatment. Systemic therapy with oral study agent, nirogacestat, will be given for 3 cycles (1 cycle = 28 days) followed by a single cryoablation procedure between Cycles 3 and 4, and then continued nirogacestat for Cycles 4 through 26. Treatment with nirogacestat may continue via this study for up to 24 months (26 cycles of treatment), unless there is progression of disease, intolerance, subject withdraws their consent, start of a new anticancer therapy, or until Subject Study Completion or Termination occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically-confirmed diagnosis of desmoid tumor (DT) that is progressing (by RECIST criteria over the past 12 months) or symptomatic (as defined by change in pain regimen or impairment of activities of daily living (ADLs), or at investigator discretion). Note: Must have diagnosis of desmoid tumor on pathology report.
2. Desmoid tumor is 50 to <75% cryoablatable.

   Tumors that are 50 to <75% (volume) ablatable in a single session are characterized by:
   1. Proximity (< 1 cm) to critical structures, such as nerves, vessels, bowel, or skin, at risk of injury during ablation, despite hydrodissection
   2. Large size ( > 100 mL)
   3. Complex shape, such that parts of the tumor cannot be reached from a single approach or subject position
   4. Thin, infiltrative components, where ablation of that portion would damage more normal anatomy than tumor (e.g., tumor extending along a fascial plane between muscles, such that ablation would damage more muscle than tumor volume)
3. If participant is currently being treated with any therapy for the treatment of DT, this must be completed at least 28 days (or 5 half-lives, whichever is shorter) prior to first dose of study treatment. All toxicities from prior therapy must be resolved to ≤ Grade 1 or clinical baseline.
4. Participants who are receiving chronic nonsteroidal anti-inflammatory drugs (NSAIDs) as treatment for conditions other than DT must be on a stable dose for at least 28 days prior to first dose of study treatment.
5. Age ≥ 18 years.
6. Participant has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 at screening.
7. Participant has adequate organ and bone marrow function as defined by the following screening laboratory values:

   1. Absolute neutrophil count ≥ 1500 cells/μL;
   2. Platelets ≥ 100,000μL;
   3. Hemoglobin ≥ 9 g/dL;
   4. Total bilirubin ≤ 1.5 × upper limit of normal (ULN) (isolated bilirubin > 1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%);
   5. Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase)/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase) ≤ 2 × ULN; and
   6. Serum creatinine ≤ 1.5 × ULN or if creatinine > 1.5 × ULN then calculated creatinine clearance must be ≥ 60 mL/min (using the Cockcroft-Gault formula)
8. Women of childbearing potential must have a negative serum pregnancy test at screening.
9. Participant can swallow tablets.
10. Participant able to have MRI.
11. Ability to understand and the willingness to personally sign the written IRB-approved informed consent document.
12. Contraceptive use by men or women should be consistent with the standard that will be used at Stanford regarding the methods of contraception for those participating in clinical studies.

    1. Male participants: Male participants are eligible to participate if they agree to the following during the treatment period and for at least 90 days after the last dose of study treatment:

       • Refrain from donating or preserving sperm;

       PLUS either:
       * Be abstinent from sexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent; OR
       * Must agree to use a male condom when having sexual intercourse with women of childbearing potential (WOCBP). An additional form of contraception as described in Appendix G should also be used by the female partner, if she is of childbearing potential.

       Postmenopausal state (not of childbearing potential) is defined as no menses for 12 months without an alternative medical cause.
    2. Female participants: A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

       * Is not of childbearing potential (not WOCBP). OR
       * Is of childbearing potential but is abstinent or using 1 highly effective contraceptive method, as described in Appendix H during the treatment periodand for at least

         1 week after the last dose of active study treatment. A second method of contraception is required if the participant is using hormonal contraception, as coadministration with nirogacestat may alter the plasma concentrations of hormonal contraceptives resulting reduced efficacy. Additionally, the participant agrees not to harvest or donate eggs (ova, oocytes) for the purpose of reproduction during the treatment period and for at least 6 months after the last dose of active study treatment. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study treatment.
       * The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.

Exclusion Criteria:

1. Participant previously received or is currently receiving therapy with GS inhibitors or anti-Notch antibody therapy.
2. Participant is currently using any treatment for DT including tyrosine kinase inhibitors (TKIs), NSAIDS (chronic daily use - except as in inclusion criterion 4) or any investigational treatment 28 days (or 5 half-lives, whichever is longer) prior to the first dose of study treatment.
3. Participant is currently using or anticipates using food or drugs that are known strong or moderate cytochrome P450 3A4 (CYP3A4) inhibitors, or strong CYP3a inducers within 14 days prior to the first dose of study treatment.
4. Participant has known hypersensitivity to the active substance or to any of the excipients of nirogacestat.
5. Participant with active or chronic infection at the time of informed consent and during the screening period.
6. Participant has known malabsorption syndrome or preexisting gastrointestinal condition that may impair absorption of nirogacestat (e.g., gastric bypass, lap band, or other gastric procedures that would alter absorption); delivery of nirogacestat via nasogastric tube or gastrostomy tube is not allowed.
7. History of other high-grade malignancy ≤ 2 years previous. Exceptions include prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen; adequately treated basal cell or squamous cell skin cancer; or adequately treated, with curative intent, cancer from which the subject is currently in complete remission per study Principal Investigator's (PI's) judgment. Specific situations can be discussed with study PI.
8. Participant has experienced any of the following within 6 months of signing informed consent:

   * Clinically significant cardiac disease (New York Heart Association Class III or IV);
   * Myocardial infarction
   * Severe / unstable angina
   * Coronary / peripheral artery bypass graft
   * Symptomatic congestive heart failure
   * Cerebrovascular accident
   * Transient ischemic attack
   * Symptomatic pulmonary embolism
9. Participant has congenital long QT syndrome.
10. Participant has a history of additional risk factors for Torsades de pointes (TdP) (e.g., heart failure, hypokalemia, family history of long QT syndrome).
11. Participant has current or chronic history of liver disease or known hepatic or biliary abnormalities (except for Gilbert's syndrome or asymptomatic gallstones).
12. Participant is currently enrolled or was enrolled within 28 days of first dose of study treatment in another clinical study with any investigational drug or device.

All subject files must include supporting documentation to confirm subject eligibility. The method of confirmation can include, but is not limited to, laboratory test results, radiology test results, subject self-report, and medical record review.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit per RECIST v1.1 | 1 year
  Clinical benefit (CB) is defined as the number of participants assessed with a complete response (CR), partial response (PR), or stable disease (SD) within 1 year and with no evidence of loss of response nor progression within that year. Response & progression will be assessed according to the Revised Response Evaluation Criteria in Solid Tumors (RECIST)v1.1, as follows:
  RECIST v1.1:
  * CR=Disappearance of all lesions
  * PR=≥30% decrease in diameter of target lesions
  * Progressive disease (PD)=20% increase in diameter of target lesion; progression of non-target lesion; or ≥1 new lesion(s)
  For the overall outcome:
  * SD=Changes not meeting above criteria
  * Overall Response (OR)=CR+PR
  * CB=CR+PR+SD

SECONDARY OUTCOMES:
Clinical Benefit per mRECIST | 1 year
  Clinical benefit (CB) is defined as the number of participants assessed with a complete response (CR), partial response (PR), or stable disease (SD) within
  1 year and with no evidence of loss of response nor progression within that year.
  Response & progression will be assessed according to the modified Revised Response Evaluation Criteria in Solid Tumors (mRECIST), as follows.
  CR=Disappearance of intratumoral enhancement
  * PR=≥ 30% decrease in the diameter of target lesion(s)
  * PD=An increase of >20% in the diameter of target lesion. The outcome is the number of participants alive after 1 year and without PD per mRECIST, a number without dispersion
Progression-free Survival (PFS) | 1 year
  Progressive-free survival (PFS) is an assessment of the number of participants at a specific time who remain alive and without tumor progression. Progressive disease (PD) will be assessed according to Revised Response Evaluation Criteria in Solid Tumors (RECIST)v1.1, or, for tumors assessed with MRI enhancement, modified RECIST (mRECIST) defined as follows:
  RECIST v1.1:
  * PD=20% increase in diameter of target lesion; progression of non-target lesion; or ≥1 new lesion(s) mRECIST:
  * PD=An increase of >20% in the diameter of target lesion. The outcome is the number of participants alive after 1 year and without PD per RECIST or mRECIST, a number without dispersion.
Objective Response | 1 year
  Objective response (OR) is defined as the number of participants assessed with a complete response (CR) or partial response (PR) within 1 year and with no evidence of loss of response nor progression within that year. Response & progression will be assessed according to the Revised Response Evaluation Criteria in Solid Tumors (RECIST)v1.1, or, for assessed with MRI enhancement, modified RECIST (mRECIST).
Time-to-Response (TTR) | 1 year
  Time-to-response (TTR) is an assessment of the length of time from the start of treatment until clinical response (complete response, CR; or partial response, PR) is documented.in accordance with the Revised Response Evaluation Criteria in Solid Tumors (RECIST)v1.1, or, for assessed with MRI enhancement, modified RECIST (mRECIST) defined as follows:'
  RECIST v1.1:
  * CR=Disappearance of all lesions
  * PR=≥30% decrease in diameter of target lesions Progressive disease (PD)=20% increase in diameter of target lesion; progression of non-target lesion; or ≥1 new lesion(s) mRECIST:
  * CR=Disappearance of intratumoral enhancement
  * PR=≥ 30% decrease in the diameter of target lesion(s) PD=An increase of >20% in the diameter of target lesion.
  For either:
  • SD=Changes not meeting above criteria The outcome is expressed as the median TTR (by RECIST or mRECIST), with standard deviation.
Duration of Response (DoR) | 1 year
  Duration of response (DoR) is defined as the time from the date of documented disease response (complete response, CR; or partial response, PR) to the date of the first documented disease progression. CR and PR will be assessed according to the Revised Response Evaluation Criteria in Solid Tumors (RECIST)v1.1, or, for assessed with MRI enhancement, modified RECIST (mRECIST) as RECIST v1.1.
Related Adverse Events (AEs) | 1 year
  Safety is assessed as the number of adverse events determined by the investigator to be possibly, probably, or definitely related to nirogacestat treatment (ie, drug toxicities). All related events will be collected and reported. Adverse events of Grade 3 (severe) are considered notable and potentially actionable during treatment, while adverse events Grade 1 or 2 are considered routine, with typically little or no change in treatment needed. The outcome will be reported as the number of related adverse events Grade 3 or higher is a number without dispersion.

CONTACTS AND LOCATIONS:
Overall Officials: Nam Bui, M.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT05949099/Prot_002.pdf